CLINICAL TRIAL: NCT01850628
Title: NSABP Biospecimen Discovery Project
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Breast Cancer Research Foundation (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NSABP DP-1
Record Dates: First submitted 2013-05-01; First posted 2013-05-09 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: National Surgical Adjuvant Breast and Bowel Project (NSABP); paclitaxel; trastuzumab; pertuzumab; HER2 positive (human epidermal growth factor receptor 2); Proteomics; Neoadjuvant Therapy; Anthracycline therapy; Locally advanced; Operable; Biomarkers
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; pertuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh tumor tissue and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paclitaxel plus trastuzumab or trastuzumab/pertuzumab: Patient received paclitaxel plus trastuzumab or a trastuzumab/pertuzumab-based combination administered per investigators discretion
  Interventions: Drug: Paclitaxel; Biological: trastuzumab; Biological: pertuzumab

INTERVENTIONS:
Drug: Paclitaxel
Biological: trastuzumab
  Other Names: Herceptin
Biological: pertuzumab

SUMMARY:
This study is a biospecimen discovery project that will serve as a pilot for a comprehensive 'omics approach using fresh core biopsy tissue and blood samples for DNA and protein analysis, as well as paired tumor-normal exome DNA and RNA sequencing.

DETAILED DESCRIPTION:
This study will be conducted at select NSABP sites where investigators are willing to give paclitaxel plus trastuzumab or a trastuzumab/pertuzumab-based combination as the initial component of neoadjuvant therapy as a pilot for a comprehensive 'omics approach using next generation sequencing and protein expression and post-translational modification analysis using mass spectrometry (MS) based and Reverse Phase Protein Array-based proteomics. Tumor samples will be obtained at baseline and 48 to 72 hours after initial drug treatment to study variation in the biological responses to these agents. The study of tumors both before and early after the first treatment probes the biological responses to treatment and is rich source of predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy or limited incisional biopsy.
* The breast cancer must be HER2-positive based on current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) Guideline Recommendations for Human Epidermal Growth Factor Receptor 2 Testing in Breast Cancer.
* The patient must have a mass in the breast measuring greater than or equal to 2.0 cm by physical exam and/or ultrasound that is accessible and safe for repeat biopsy. Patients with a diagnosis of inflammatory breast cancer are eligible if there is a palpable or detectable breast mass that is accessible and safe for repeat biopsy.
* Planned initial treatment with a combination of paclitaxel and trastuzumab or a trastuzumab/pertuzumab-based combination. Schedule for paclitaxel/trastuzumab or trastuzumab/pertuzumab administration is per the investigator.

Exclusion Criteria:

* Excisional biopsy or lumpectomy performed prior to registration.
* Previous therapy with chemotherapy or targeted therapy for any malignancy.
* Treatment, including radiation therapy (RT), chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to registration.
* Other nonmalignant systemic disease that would preclude the patient from receiving chemotherapy and targeted therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with locally advanced, HER2-positive breast cancer from selected sites in the United States
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-06 (Actual); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Measure variation in biologic response by comprehensive tumor 'omics profiling in patients receiving an upfront regimen containing paclitaxel plus trastuzumab or a trastuzumab/pertuzumab-based combination | blood and tissue specimens will be collected at the time of diagnosis; prior to treatment; 48 and 72 hours following first dose of treatment; and following surgery, if tumor remains.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas